CLINICAL TRIAL: NCT03653065
Title: Assiut University Children Hospital
Brief Title: Assiut University Children Hospital Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, nora hassan, principle investigator, Assiut University
Other Study IDs: Mechanical ventilation
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Ventilation Outcomes

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frequency and outcomes of mechanical ventilation In intensive care unit at Assiut university children hospital.

DETAILED DESCRIPTION:
Data will be extracted from the files of the patients which will include the following:

History Examination Investigations Cause of mechanical ventilation (status epilepticus,respiratory failure and other) First attempt success rate

ELIGIBILITY:
Inclusion Criteria:

* Patients who are mechanically ventilated
* age:One month to 18 years.
* sex:both male and female
* duration:for one year
* type of the study:retrospective
* site :intensive care unit at Assiut university children hospital

Exclusion Criteria:

* patients who are intubated outside Assiut university children hospital.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Data will be extracted from the files of the patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of endotracheal intubation | one year
  will be calculated by the following equiation : Number of patient who undergo endotracheal intubation over total number of patient admitted to intensive care unit × 100 .
First attempt success rate | one year
  will be calculated by comparing the number of patients on whom ETI was attempted with the times successful tracheal intubation was achieved on a first attempt at laryngoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nora, Asyut, Egypt